CLINICAL TRIAL: NCT06491446
Title: A Randomized, Placebo-Controlled Study to Evaluate Clearance of High-Risk Human Papillomavirus and Safety After Administration of ABI-2280 Vaginal Inserts
Brief Title: Evaluating Clearance of High-Risk HPV and Safety After Administration of ABI-2280 Vaginal Inserts
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antiva Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-2280-401
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV; sexually-transmitted infection; high-risk HPV; CIN
MeSH Terms: conditions — Papillomavirus Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Experimental: Cohort 1 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 1) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 2 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 2) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 3 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 3) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 4 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 4) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 5 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 5) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 6 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 6) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 7 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 7) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 8 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 8) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 9 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 9) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 10 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 10) or matching placebo
  Interventions: Drug: ABI-2280
- Experimental: Cohort 11 (Active Comparator): Participants in this arm will receive either ABI 2280 (Dose 11) or matching placebo
  Interventions: Drug: ABI-2280

INTERVENTIONS:
Drug: ABI-2280 — Different strength of ABI 2280 will be administered in different cohorts.
  Other: Placebo Matching placebo will be administered.

SUMMARY:
This is a blinded study to assess safety, tolerability, and efficacy of ABI-2280 vaginal inserts in participants diagnosed with persistent cervical hrHPV infection. This study will have up to 11 cohorts with various dose strengths and regimens. Each cohort will start with a sentinel cohort of 8 participants. Sentinel cohorts may be expanded to include an additional up to 32 participants to provide additional proof of concept data to further understanding of benefit/risk of a given dose/dose regimen.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 1b/2 study in women diagnosed with persistent cervical hrHPV infection. This study is designed to assess safety, tolerability, and efficacy following the use of ABI-2280 Vaginal Insert delivered intravaginally. Sentinel cohorts will be utilized to assess tolerable regimens, which may trigger cohort expansions if some evidence of efficacy is observed.

Dose range and dosing regimens in this study will be evaluated through the enrollment of up to 11 sentinel cohorts, each enrolling up to 8 participants.

ELIGIBILITY:
Inclusion Criteria

* Female sex, 25 to 55 years of age
* Positive hrHPV result on at least 2 consecutive tests prior to randomization, one hrHPV+ result at least 12 months prior to screening
* Cervical cytology, colposcopy and/or biopsy performed within the last 6 months confirming disease status no greater than low-grade squamous intraepithelial lesions or cervical intraepithelial neoplasia grade 1.

Exclusion Criteria

* History of biopsy or colposcopy indicating high-grade squamous intraepithelial lesions, or history of endocervical curettage positive for glandular dysplasia
* Any clinically significant immune suppressing condition
* History or current diagnosis of cervical cancer, suspected or confirmed
* Plan to have excision or ablation of cervical or vaginal lesions, or to undergo large loop excision of the transformation zone at any time during the study.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
For sentinel cohorts: Incidence and Severity of Adverse Events | Week 24
  For sentinel cohorts: for each dose/dosing regimen, incidence and severity of adverse events (AEs), relationship of AEs to investigational product (IP), and AEs leading to treatment reduction/discontinuation for ABI-2280 Vaginal Insert vs. pooled placebo
For fully expanded cohorts, including sentinel: Clearance of persistent cervical hrHPV infection as defined by the absence of all hrHPV genotypes present at baseline | Week 12
  Proportion of participants who received ABI-2280 vs pooled placebo who are complete responders.

SECONDARY OUTCOMES:
For fully expanded cohorts, including sentinel: Incidence and Severity of Adverse Events | Week 24
  For fully expanded cohorts, including sentinel: for each dose/dosing regimen, incidence and severity of AEs, relationship of AEs to IP, and AEs leading to treatment reduction/discontinuation for ABI-2280 Vaginal Insert vs. pooled placebo.
Proportion of participants who received ABI-2280 vs pooled placebo who are complete responders | Week 24
  For fully expanded cohorts, including sentinel: For each dose/dosing regimen, proportion of participants who received ABI-2280 Vaginal Insert vs. pooled placebo who are complete responders, defined as the absence of all hrHPV genotypes that were present at baseline, at Week 24

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (8):
  - PARC Clinical Research, Royal Adelaide Hospital, Adelaide, South Australia
  - Emeritus Research Camberwell, Camberwell
  - Holdsworth House Medical Practice, Darlinghurst
  - KIMR, Nedlands
  - The Royal Women's Hospital, Parkville
  - Emeritus Research Sydney, Sydney
  - AusTrials Taringa, Taringa
  - AusTrials Wellers Hill, Tarragindi
- New Zealand (8):
  - Waitemata Clinical Research Ltd, Birkenhead
  - P3 Research Dunedin, Dunedin
  - P3 Research Hawke's Bay, Hastings
  - P3 Research Lower Hutt, Lower Hutt
  - Pacific Clinical Trials Network - Tasman, Nelson
  - P3 Research Kapiti, Paraparaumu
  - Lakeland Clinical Trials, Rotorua
  - Clinical Horizons New Zealand, Tauranga